CLINICAL TRIAL: NCT05392920
Title: Determination of the Validity of One-Minute Sit-to-Stand Test in Obese and Overweight Children and Adolescents
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, nesrine benkhalifa, Principal Investigator, Istanbul University - Cerrahpasa
Other Study IDs: 2022/37
Record Dates: First submitted 2022-05-15; First posted 2022-05-26 (Actual); Last update posted 2022-07-08 (Actual); Status verified 2022-07

CONDITIONS: Obese; Child Obesity; Adolescent Obesity; Exercise Capacity
Keywords: obese patient; functional test; reliability; validity
MeSH Terms: conditions — Obesity; Pediatric Obesity | interventions — Outcome Assessment, Health Care

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Obese children and adolescents: Obese children and adolescent patients
  Interventions: Other: assessment study

INTERVENTIONS:
Other: assessment study — there is no intervention in this study

SUMMARY:
Obese individuals need to be evaluated comprehensively before exercise programs are determined. Determination of exercise intolerance is important for the detection of functional limitations. One minute sit to stand test (1MSTST) can be used as an alternative to cardiopulmonary exercise tests (CPET) or field tests. It is easy to use, quick to apply, valid and reliable, and applicable even in small areas. In addition, it is a simple assessment adequate for children's needs and behaviors and can be easily applied both in the clinic and at home, making it easier to use in children. Studies have shown that 1MSTST is a valid test in chronic obstructive pulmonary disease (COPD), cystic fibrosis, interstitial lung disease, and, healthy children and adolescents. However, no study has been found regarding the validity of its use in obese children and adolescents.The aim of our study is to investigate the validity and reliability of 1MSTST in overweight-obese children and adolescents.

ELIGIBILITY:
Inclusion Criteria:

* Being in the 8-18 age range.
* Being overweight (between 85 and 95 according to the Body Mass Index percentile).
* Being obese (over 95 based on the Body Mass Index percentile).
* Not doing any vigorous exercise two hours before the test.

Exclusion Criteria:

* History of hospitalization in the last month for a reason that may affect physical performance.
* Having neurological, musculoskeletal disease that prevents exercise tests.
* Uncontrollable medical conditions (Cardiovascular, pulmonary disease, etc.).
* Visual and/or vestibular disorders.

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Overweight or obese children and adolescents
Sampling Method: Non-Probability Sample
Enrollment: 28 (Estimated)
Dates: Start 2022-07-08 (Estimated); Primary Completion 2022-10-02 (Estimated); Study Completion 2022-11-02 (Estimated)

PRIMARY OUTCOMES:
1 min sit to stand test | Baseline
  Only a chair and a stopwatch are needed to apply the test. It is recommended to use a chair with a height of 45-48 cm, preferably against the wall, fixed, without arm support. The patients will sit with their feet flat on the ground and cross their arms over the chest. The patient will be asked to get up from the chair and sit down as fast as he/she can for 1 minute. The number of standing up will be recorded.
6 minute walk test | Baseline
  The patient's exercise capacity will be determined by the six minute walk test. The test will be applied in a corridor 30 meters long. The patient will be asked to walk as fast as possible for six minutes. The patient can stop during the test if they needed. The total time, the number of times it has stopped and the total distance traveled will be recorded. Oxygen saturation, heart rate, and blood pressure measurements will be taken before and after the test. According to the modified Borg scale, dyspnea, leg fatigue and general fatigue will be questioned.

SECONDARY OUTCOMES:
Waist circumference | Baseline
  Waist circumference will be measured using a tape measure from the midpoint between the lowest rib and the iliac crest, when the patient is standing .
Hip circumference | Baseline
  Hip circumference will be measured parallel to the ground with a tape measure at the level of the trochanter major.
Body fat percentage | Baseline
  Body fat percentage will be analyzed with the BIA instrument (Tanita MC 780 MA Body Composition Analysis, Amsterdam, Netherlands).
Body muscle percentage | Baseline
  Body muscle percentage will be analyzed with the BIA instrument (Tanita MC 780 MA Body Composition Analysis, Amsterdam, Netherlands).

CONTACTS AND LOCATIONS:
Overall Officials: Goksen Kuran Aslan, PT, phD, Study Director — Istanbul University - Cerrahpasa
Locations (1):
- Istanbul University-Cerrahpasa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bohannon RW, Crouch R. 1-Minute Sit-to-Stand Test: SYSTEMATIC REVIEW OF PROCEDURES, PERFORMANCE, AND CLINIMETRIC PROPERTIES. J Cardiopulm Rehabil Prev. 2019 Jan;39(1):2-8. doi: 10.1097/HCR.0000000000000336. PMID 30489442
- [Background] ATS Committee on Proficiency Standards for Clinical Pulmonary Function Laboratories. ATS statement: guidelines for the six-minute walk test. Am J Respir Crit Care Med. 2002 Jul 1;166(1):111-7. doi: 10.1164/ajrccm.166.1.at1102. No abstract available. PMID 12091180
- [Background] Ozgen IT, Cakir E, Torun E, Gules A, Hepokur MN, Cesur Y. Relationship Between Functional Exercise Capacity and Lung Functions in Obese Chidren. J Clin Res Pediatr Endocrinol. 2015 Sep;7(3):217-21. doi: 10.4274/jcrpe.1990. PMID 26831556
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/30489442/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/12091180/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/26831556/